CLINICAL TRIAL: NCT07043699
Title: Effect of Phonophoresis Versus Iontophoresis in the Treatment of Perimenopausal Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mereet Mokhles Zaref Farid, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005763
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Phonophoresis; Iontophoresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phonophoresis (Experimental): It consisted of 21 perimenopausal women. Each patient in this group received phonophoresis, 3 times per week, for 8 weeks.
  Interventions: Other: Phonophoresis
- Iontophoresis (Experimental): It consisted of 21 perimenopausal women. Each patient in this group received iontophoresis, 3 times per week, for 8 weeks.
  Interventions: Other: Iontophoresis

INTERVENTIONS:
Other: Phonophoresis — Each woman in the first group received phonophoresis treatment. The procedure was performed using diclofenac sodium gel. Treatment was administered three times per week over a period of eight weeks. Ultrasound was applied at an intensity of 1 W/cm² for 8 minutes using a pulsed mode at a frequency of 1 MHz.
  Arms: Phonophoresis
Other: Iontophoresis — Each woman in the second group received iontophoresis treatment using a diclofenac sodium solution (Voltaren ampoules). The solution was applied under the cathode (drug delivery electrode). The iontophoresis leads were connected, and the current intensity was adjusted based on individual tolerance, ranging between 1 and 4 mA, for a duration of 20 minutes. The negative electrode was placed on the medial side of the calcaneal tubercle (origin), while the positive electrode was positioned on the forefoot. Treatment was administered three times per week over a period of eight weeks.
  Arms: Iontophoresis

SUMMARY:
The purpose of the study was to investigate the effect of phonophoresis versus iontophoresis on plantar fasciitis in perimenopausal women.

DETAILED DESCRIPTION:
Collagen plays a critical role in determining the tensile strength of connective tissue. During the perimenopausal transition, the overall quantity of collagen decreases; however, there is a relative increase in type I collagen compared to type III collagen. This shift contributes to increased tissue stiffness. Research indicates that estrogen has a protective effect on muscles and fascia, preventing fibrogenesis. Consequently, as estrogen levels decline during perimenopause, fibrogenic activity may increase. In addition, reduced estrogen levels are associated with enhanced elastin degradation, leading to diminished tissue elasticity and reduced recoil capacity.

This degradation of connective tissue is considered a primary cause of plantar fasciitis, which results from collagen breakdown in the plantar fascia at its origin-the calcaneal tuberosity of the heel-and surrounding fascial structures.

When plantar fasciitis develops in perimenopausal women, it can significantly disrupt daily activities. Many women experience fallen arches and severe irritation, with pain affecting functions such as standing, walking, climbing stairs, and working. This functional impairment can lead to emotional consequences, including depression.

Given these challenges, there is a pressing need to identify new, alternative, and cost-effective methods for managing and treating this condition. This study examined the effectiveness of phonophoresis and iontophoresis in treating plantar fasciitis in perimenopausal women. The findings aimed to contribute valuable knowledge to the field of physical therapy and offer practical solutions for women suffering from this condition.

ELIGIBILITY:
Inclusion Criteria:

* All participants were perimenopausal women who had been suffering from plantar fasciitis (PF) for at least one month.
* Patients reported heel pain during the first step in the morning, while bearing weight, and after walking or running.
* Diagnosis was confirmed using the Windlass test, Tarsal Tunnel test, and tenderness at the anterior medial heel.
* Participants were aged between 50 and 51 years and experienced menstrual irregularities.
* Their body mass index (BMI) was greater than 30 kg/m².
* They had not received any medical treatment for plantar fascia pain or collagen supplements.
* None of the participants were on hormonal therapy.

Exclusion Criteria:

* Patients with a history of rheumatoid arthritis, diabetes mellitus, or hypertension.
* Those diagnosed with neurological disorders.
* Individuals who had undergone previous foot surgeries, experienced burns, or suffered severe foot trauma.
* Participation in any other exercise training program during the study period.
* History of skeletal deformities.
* Presence of knee or ankle replacements.
* Presence of ankle plates, screws, or nails.
* Notable differences in lower limb length.
* History of foot fractures that resulted in deformities.
* Presence of infective foot conditions, dermatitis, or tumors.
* Impaired circulation in the lower extremities.
* Corticosteroid injection to the heel within the past year.
* Congenital foot deformities.

Ages: 50 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Assessment of pain | 8 weeks
  The Visual Analog Scale (VAS) was used to assess pain levels in each woman in both groups before and after the treatment program. Pain scores were determined by measuring the distance in millimeters on a 10-cm line between the "no pain" anchor and the patient's mark, yielding a score from 0 to 100. Higher scores indicated greater pain intensity. Recommended cut points were: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

SECONDARY OUTCOMES:
Measurement of the level of disability | 8 weeks
  Foot function was measured before and after the treatment program using the Foot Function Index (FFI), a self-reported, foot-specific tool used for over 20 years to assess pain and disability. The FFI consisted of 23 items divided into three subscales: pain, disability, and activity limitation. Scores were interpreted on a scale from 0% to 100% for each subscale and for the overall index. Higher scores indicated poorer foot health and reduced foot-related quality of life.
Assessment of Dorsi flexion Range of Motion (ROM) | 8 weeks
  Dorsiflexion ROM was measured using an inclinometer placed at the tibial tuberosity and distal tibia. Participants performed a knee-bent stance facing a wall, with the dominant foot stepped back and toes forward. They bent the dominant knee forward while keeping the foot flat and used the wall for balance if needed. The examiner measured dorsiflexion once full foot contact could no longer be maintained. The inclinometer was calibrated before each session, and values were recorded to the nearest degree. Three consistent trials within ±5° or ±10% were required, with up to six attempts allowed.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Mohamed Hanfi Emara, PhD, Study Chair — Professor, Cairo university; Hossam Eldin Hossam Eldin Hussein Kamel, PhD, Study Director — Professor, Al-Azhar university
Locations (1):
- Cairo University, Giza, Egypt